CLINICAL TRIAL: NCT07283666
Title: Subspecialty Ambulatory Quality Cardiology Program: An Audit and Feedback Performance Improvement Strategy
Brief Title: Subspecialty Ambulatory Quality Cardiology Program
Status: Enrolling by invitation | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-Specialty Ambulatory
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quarterly Emails: Quarterly emails on performance will be sent.
- Control: Usual Care (no emails on performance).

SUMMARY:
Investigators will evaluate the effectiveness of an audit and feedback performance improvement strategy in which cardiology providers receive quarterly emails on ambulatory quality improvement goals.

ELIGIBILITY:
Inclusion Criteria for atrial fibrillation quality metric:

* Active diagnosis of atrial fibrillation
* CHADS2VASC of at least 2 in males and at least 3 in females
* Outpatient cardiology visit in past 3 months

Inclusion Criteria for HFrEF quality metric:

* Most recent EF ≤40
* Age 18-90
* Outpatient cardiology visit in past 3 months

Exclusion Criteria for atrial fibrillation quality metric:

* LAAO device
* Hemorrhagic Stroke

Exclusion Criteria for HFrEF quality metric:

* SBP<90
* eGFR<30
* Potassium>5
* Active allergy to MRA
* Acknowledge reason on heart failure alert
* Mechanical circulatory device
* Cardiac amyloid diagnosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen by a cardiology provider in the ambulatory setting.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients eligible for medications who are prescribed these medications | Day 1

SECONDARY OUTCOMES:
Percentage of patients with HFrEF prescribed aldosterone antagonists | Day 1
Percentage of patients with Afib prescribed oral anticoagulants | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Mukhopadhyay, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a quality improvement (QI) project and individual participant data (IPD) will not be shared with other researchers.